CLINICAL TRIAL: NCT00002389
Title: A Randomized, Double-Blind, Parallel-Group, Multicenter Trial to Evaluate the Safety and Efficacy of 1592U89 in Combination With Lamivudine (3TC) and Zidovudine (ZDV) Versus 3TC/ZDV in HIV-1-Infected, Antiretroviral Therapy-Naive Subjects With CD4+ Counts >= 100 Cells/mm3
Brief Title: The Safety and Effectiveness of Lamivudine Plus Zidovudine, Used With and Without 1592U89, in HIV-1 Infected Patients Who Have Never Taken Anti-HIV Drugs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Model: Parallel | Purpose: Treatment
Other Study IDs: 238D
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-11

CONDITIONS: HIV Infections
Keywords: HIV-1; Drug Therapy, Combination; Antiviral Agents; Zidovudine; CD4 Lymphocyte Count; Lamivudine; RNA, Viral; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load; abacavir
MeSH Terms: conditions — HIV Infections | interventions — abacavir; Lamivudine; Zidovudine

INTERVENTIONS:
Drug: Abacavir sulfate
Drug: Lamivudine
Drug: Zidovudine

SUMMARY:
To compare the durability of the viral load response following 48 weeks of treatment with 1592U89/lamivudine (3TC)/zidovudine (ZDV) versus 3TC/ZDV alone. To compare the early antiviral activity following 16 weeks treatment with 1592U89/3TC/ZDV versus 3TC/ZDV alone as demonstrated by the proportion of subjects with viral load < 400 copies/ml, plasma HIV-1 RNA profiles and CD4+ profiles. To assess the safety and tolerance following 16 and 48 weeks of treatment with 1592U89/3TC/ZDV versus 3TC/ZDV alone.

DETAILED DESCRIPTION:
This study compares the safety and efficacy of 1592U89 in combination with 3TC and ZDV versus control therapy with 3TC and ZDV alone. If a patient has two consecutive HIV-1 RNA measurements of >= 400 copies/ml (performed at least one week apart) he or she has the option to switch to open-label therapy with 1592U89/3TC/ZDV, to receive the remaining randomized treatment, or to discontinue study medication. If this criterion is not met, patients continue their randomly assigned therapy until the last patient has completed 48 weeks of therapy. Once patients enter the open-label phase, investigators may add or substitute non-nucleoside reverse transcriptase inhibitors, nucleoside reverse transcriptase inhibitors, or protease inhibitors for 3TC and/or ZDV according to their standard practice once patients enter the open-label phase.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Local treatment for Kaposi's sarcoma.
* Hematologic supportive therapy with GM-CSF, G-CSF, or erythropoietin.

Patients must have:

* HIV-1 infection as documented by a licensed HIV-1 antibody ELISA and confirmed by either Western blot detection of HIV-1 antibody or positive HIV-1 blood culture.
* One screening CD4 lymphocyte cell count >= 100 cells/mm3 within 14 days prior to study drug administration.
* No active or ongoing AIDS-defining opportunistic infection or disease.
* Signed, informed consent from parent or legal guardian for patients under 18 years of age.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions and symptoms are excluded:

* Malabsorption syndrome or other gastrointestinal dysfunction that might interfere with drug absorption or render the patient unable to take oral medication.
* Serious medical conditions such as diabetes, congestive heart failure, cardiomyopathy, or other cardiac dysfunction, that, in the opinion of the investigator, would compromise the safety of the patient.

Concurrent Medication:

Excluded:

* Foscarnet therapy.
* Immunomodulating agents such as systemic corticosteroids, interleukins, thalidomide, anti-cytokine agents, or interferons.
* Cytotoxic chemotherapeutic agents and antioxidants.

Concurrent Treatment:

Excluded:

Radiation therapy.

Patients with the following prior conditions are excluded:

History of clinically relevant pancreatitis or hepatitis within the last 6 months.

Prior Medication:

Excluded:

* Prior antiretroviral therapy.
* Vaccination within the past 3 months given as part of an investigational HIV vaccine trial.
* Chemotherapeutic agents within 30 days of study drug administration.
* Immunomodulating agents such as systemic corticosteroids, interleukins or interferons, within 30 days of study drug administration.

Prior Treatment:

Excluded:

Radiation therapy within 30 days of study period. Current alcohol or illicit drug use that, in the opinion of the investigator, may interfere with the patient's ability to comply with the dosing schedule and protocol evaluations.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 210

CONTACTS AND LOCATIONS:
Locations (15):
- United States (13):
  - East Bay AIDS Ctr, Berkeley, California
  - Kraus Med Partners, Los Angeles, California
  - Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - Univ of Miami Dept of Medicine, Miami, Florida
  - Rush Med College / Rush Presbyterian - St Luke's Med Cen, Chicago, Illinois
  - Boston Med Ctr / Evans - 556, Boston, Massachusetts
  - Saint Michael's Med Ctr / Dept of Infectious Diseases, Newark, New Jersey
  - St Vincent's Hosp and Med Ctr / AIDS Ctr, New York, New York
  - Harlem Hosp, New York, New York
  - Duke Univ Med Ctr / Dept of Medicine, Durham, North Carolina
  - Univ of Cincinnati / Holmes Hosp, Cincinnati, Ohio
  - Dr Nicholaos Bellos, Dallas, Texas
  - Baylor College of Medicine / Dept of Medicine, Houston, Texas
- Toronto Gen Hosp, Toronto, Ontario, Canada
- San Juan AIDS Program, Santurce, Puerto Rico